CLINICAL TRIAL: NCT04733768
Title: 18F-PSMA-1007 PET/CT Imaging in Patients with Biochemically Recurrent or High-risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CC-20-0281
Record Dates: First submitted 2020-12-11; First posted 2021-02-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-PSMA-1007 PET/CT scan (Experimental): Single Arm study - all enrolled patients will undergo an experimental 18F-PSMA-1007 PET/CT scan
  Interventions: Diagnostic Test: 18F-PSMA-1007

INTERVENTIONS:
Diagnostic Test: 18F-PSMA-1007 — 18f-PSMA-1007 PET/CT scan
  Other Names: [18F]PSMA-1007

SUMMARY:
Single centre prospective cohort phase II study of 18F-PSMA-1007 PET/CT imaging in patients with biochemically recurrent or high-risk prostate cancer. Safety, biodistribution, clinical efficacy, and diagnostic accuracy will be assessed. For diagnostic accuracy comparison will be made to a contemporary (within 10 days) conventional imaging study (bone scan and CT scan).

DETAILED DESCRIPTION:
A single centre prospective cohort phase II study of 18F-PSMA-1007 PET/CT imaging in specific patient populations:

1. Adult patients (≥ 18 years old) with a history of radical prostatectomy for treatment of prostate cancer, and a serum prostate specific antigen (PSA) > 0.2 µg/L
2. Adult patients (≥ 18 years old) with a history of radiotherapy, cryotherapy, or brachytherapy for treatment of prostate cancer, and a serum PSA progressively rising to ≥ 2 µg/L (minimum two samples) OR a serum PSA doubling-time of < 9 months
3. Adult patients (≥ 18 years old) with a history of biopsy-proven prostate cancer and high-risk features for metastatic disease prior to treatment with radical prostatectomy, radiotherapy, cryotherapy, or brachytherapy. High-risk features include a Gleason score > 7, serum PSA > 20 µg/L, OR minimum clinical T-stage T2c.

All patients will have a comparison conventional imaging study performed within 10 days of the investigational PET/CT scan. The conventional imaging study will include a 99mTc -MDP bone scan including whole body planar imaging (top of skull to toes) as well as SPECT/CT imaging of the trunk (including clavicles to pelvis). In the absence of contraindications (renal failure with eGFR < 40 mL/min/1.73m2 or history of IV contrast allergy), all scans will include an IV-contrast enhanced CT scan of the chest, abdomen, and pelvis. In the presence of contraindications to IV contrast, a non-IV contrast enhanced CT scan of the chest, abdomen, and pelvis will be performed.

The biodistribution of 18F-PSMA-1007 produced by the Edmonton PET Centre will be evaluated in 2 ways:

* by comparing the biodistribution of tracer on the scans to an expected normal distribution.
* for any identified abnormal distribution, a lesion-by-lesion comparison to the conventional imaging study will be performed with lesions classified as follows:

  * A - lesion identified on the investigational imaging study but not on the conventional imaging study
  * B - matching lesions on both the investigational and conventional imaging studies
  * C - lesion identified on the conventional imaging study but not on the investigational imaging study

The clinical efficacy of 18F-PSMA-1007 will be evaluated as follows:

• a follow-up questionnaire will be sent to referring clinicians 6 months after the scan to determine if the scans were of perceived clinical benefit.

The safety of 18F-PSMA-1007 produced by Edmonton PET Centre will be evaluated in 3 ways:

* the patients will be screened for adverse effects immediately post-injection as well as after the scan (approximately 2.5 hours after injection)
* the patients will be provided an information sheet and contact information for self-reporting of delayed adverse events (1-7 days post injection)
* a 6 month follow-up questionnaire will be sent to referring clinicians to determine if there were any perceived adverse events related to the injection

The diagnostic accuracy of 18F-PSMA-1007PET/CT produced by Edmonton PET Centre will be evaluated as follows:

* All lesions categorized as "A", "B", or "C" will be compared with a reference standard to determine sensitivity and specificity on both a per lesion and per patient level
* The reference standard will be defined a minimum of 1 year after completion of both scans based on available clinical data
* Lesional histopathology results will be used as the reference standard when available
* When pathology is unavailable, criteria for determining lesional positivity for metastatic disease will be based on recently published methodology (Lawhn-Heath et al., AJR 2019;213:1-8)
* If lesion the criteria for determining lesion positivity are not met, the lesion will be considered unevaluable and will be excluded from assessment of accuracy

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old) with a history of radical prostatectomy for treatment of prostate cancer, and a serum prostate specific antigen (PSA) > 0.2 µg/L
2. Adult patients (≥ 18 years old) with a history of radiotherapy, cryotherapy, or brachytherapy for treatment of prostate cancer, and a serum PSA progressively rising to ≥ 2 µg/L (minimum two samples) OR a serum PSA doubling-time of < 9 months
3. Adult patients (≥ 18 years old) with a history of biopsy-proven prostate cancer and high-risk features for metastatic disease prior to treatment with radical prostatectomy, radiotherapy, cryotherapy, or brachytherapy. High-risk features include a Gleason score > 7, serum PSA > 20 µg/L, OR minimum clinical T-stage T2c.

Exclusion Criteria:

1. Unable to obtain consent
2. Weight >225 kg (weight limitation of PET/CT scanner)
3. Unable to lie flat for 30 minutes to complete the PET-CT imaging session
4. Lack of intravenous access
5. Both CT scan of the chest, abdomen, and pelvis and 99mTc-MDP bone scan within 3 months
6. History of allergic reaction to 18F-PSMA-1007 or 99mTc-MDP

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Safety - immediate | Immediately (within 15 minutes) after 18F-PSMA-1007 injection
  Incidence of tracer-emergent adverse events including allergic reaction (hives, difficulty breathing) or pain at the injection site
Safety - post scan | 2.5 hours after 18F-PSMA-1007 injection
  Incidence of tracer-emergent adverse events including allergic reaction (hives, difficulty breathing) or pain at the injection site
Safety - delayed | 6 months after 18F-PSMA-1007 injection
  Questionnaire (open-ended) to referring physicians to document any perceived delayed adverse events related to 18F-PSMA-1007 tracer injection
Biodistribution | Within 5 days of scan
  Evaluation of whether tracer distribution is as expected based on published normal distribution and known disease
Diagnostic Accuracy | 1 year after 18F-PSMA-1007 PET/CT scan
  Lesion by lesion comparison to conventional imaging (bone scan and CT scan) performed 2-10 days after the 18F-PSMA-1007 PET/CT scan. Reference standard based on lesion pathology (if available) or 1 year clinical/imaging following (using criteria published by Lawhn-Heath et al., AJR 2019;213:1-8.

SECONDARY OUTCOMES:
Clinical Efficacy | 6 months after the 18F-PSMA-1007 PET/CT scan
  Questionnaire completed by referring physicians evaluating the perceived clinical effect of the 18F-PSMA-1007 PET/CT on patient management

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No